CLINICAL TRIAL: NCT06525922
Title: Center M Feasibility and Efficacy Pilot Study
Brief Title: Preventing Perinatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ellen Tilden, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OHSU IRB 24818
Record Dates: First submitted 2024-07-19; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Perinatal Depression
Keywords: Prenatal Care; Mindfulness-Based Cognitive Behavioral Therapy for Perinatal Depression; Maternal Morbidity; Maternal Mortality
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Intervention Model Description: One group was compared between pre-intervention and post-intervention time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Center M Intervention (Experimental): Data from participants in this arm will be compared across pre-intervention, post-intervention, and 6-weeks postpartum. All participants will receive the Center M intervention, which includes group-based Cognitive Behavioral Therapy (CBT) sessions and home practice materials.
  Interventions: Behavioral: Center M

INTERVENTIONS:
Behavioral: Center M — Center M consists of weekly, 1-hour, telehealth, mindfulness-based Cognitive Behavioral Therapy (CBT) group sessions for four consecutive weeks. Participants joined group sessions on their personal computer, tablet, or phone. Each visit involved the introduction of a core mental well-being theme, learning skills to develop non-judgmental self-awareness and/or cognitive reappraisal skills, skills practice, and discussion of home practice materials. Home practice materials included written mindful awareness instructions, audio-guided meditations, self-compassion exercises, and practices in recognizing the interrelationships between thoughts, feelings, and behaviors.

SUMMARY:
The goal of this pilot study is to evaluate the acceptability, feasibility, mechanisms of action, and efficacy of Center M. Center M is a group-based, mindfulness-based Cognitive Behavioral Therapy (CBT) intervention to treat Perinatal Depression (PD).

DETAILED DESCRIPTION:
The goal of this pilot study is to evaluate the acceptability, feasibility, mechanisms of action, and efficacy of Center M. Center M is a group-based, mindfulness-based Cognitive Behavioral Therapy (CBT) intervention to treat Perinatal Depression (PD). Pregnant participants will be surveyed at three time points: pre-intervention, post-intervention, and 6-weeks postpartum. Surveys will include self-report measures evaluating depressive symptoms, mindfulness skills, emotion regulation, and participant satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at intervention onset between 12 and 30 weeks
* English fluency
* no previous experience in a mindfulness-based intervention group
* ability and willingness to participate in a telehealth intervention

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | Measured at pre-intervention (within 1 week before first session), post-intervention (within 1 week after last session), and 6-weeks postpartum
  10-item self-report measure used to assess perinatal depression symptomology over the past seven days.
Patient Health Questionnaire - 8 (PHQ-8) | Measured at pre-intervention (within 1 week before first session), post-intervention (within 1 week after last session), and 6-weeks postpartum
  Self-report measure that assesses depressive symptoms over the past two weeks.
Five Facets of Mindfulness Questionnaire (FFMQ) | Measured at pre-intervention (within 1 week before first session) and 6-weeks postpartum
  39-item self-report measure to assess mindfulness skills.
Emotional Regulation Questionnaire (ERQ) | Measured at pre-intervention (within 1 week before first session) and 6-weeks postpartum
  10-item self-report measure used to assess one's ability to regulate or manage emotion using cognitive reappraisal and expressive suppression.

SECONDARY OUTCOMES:
ERQ Cognitive Reappraisal Subscale | Measured at pre-intervention (within 1 week before first session) and 6-weeks postpartum
  6 items to reflect cognitive reframing or restructuring.
ERQ Expressive Suppression Subscale | Measured at pre-intervention (within 1 week before first session) and 6-weeks postpartum
  4 items to reflect expressive suppression.
Center M Satisfaction | Post-intervention (within 1 week after last session)
  60 minute telehealth format focus groups including open-ended questions about their experience with Center M or two-question survey with a Likert scale satisfaction question and a free text question.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Tilden, PhD, CNM, FACNM, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No